CLINICAL TRIAL: NCT04018183
Title: The Role of Protein Tyrosine Kinase 7 (PTK7) in Non-small Cell Lung Cancer: Functional Analysis and Molecular Mechanism Study
Brief Title: The Role of Protein Tyrosine Kinase 7 (PTK7) in Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201902071RINC
Record Dates: First submitted 2019-05-16; First posted 2019-07-12 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-05

CONDITIONS: Tumor Progression
Keywords: non-small cell lung cancer; epidermal growth factor receptor tyrosine inhibitor
MeSH Terms: conditions — Disease Progression; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biopsy tissue, DNA, RNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To understand the mechanism and cellular functions of PTK7-associated signaling pathways in promoting lung cancer progression and conferring treatment to epidermal growth factor receptor tysosine kinase inhibitors (EGFR TKIs).

DETAILED DESCRIPTION:
* RNA extraction: We will extract total RNA from cell lysates by using Tri-reagent (Molecular Research Center, Inc., Cincinnati, Ohio) and an RNA Mini Kit (Qiagen, Hilden, Germany) according to the manufacturer's instruction. RNA obtained from the Mini Kit column will be eluted. The quantity and quality of the purified RNA will be evaluated using a NanoDrop ND-1000 spectrophotometer will be stored at -80 °C for further mutational analyses.
* Data acquisition: We will record and follow patients' clinical information, including ethnicity, age, gender, smoking status, histological types, lung cancer stage (the TNM status), metastatic sites, ECOG score, CT/CXR imaging, chemotherapy or radiation treatment at the time of diagnosis of lung cancer and through the entire clinical courses. Specific marker such as TTF1, is used to ensure the diagnosis of primary lung tumor. Clinicopathologic stage assigns according to the seventh tumor-node-metastasis classification. We assess the treatment responses according to the Response Evaluation Criteria in Solid Tumors (RECIST) using the unidimension method, and record the best response achieved per treatment. Treatment response, progression-free survival, and overall survival are recorded prospectively for further analysis.
* Statistical analysis: All categorical variables will be analyzed with Pearson's χ² test, except where a small size required the use of Fisher's exact test. The progression-free survival curve and overall survival will be plotted by the Kaplan-Meier method and compared by the log-rank test. Multivariate analysis for overall survival will be performed using the Cox's proportional hazards model. Two-sided p-values of less than 0.05 is considered significant. All analyses will be performed using SPSS software (version 16.0 for Windows; SPSS Inc.).

ELIGIBILITY:
Inclusion Criteria:

* Residual specimens under the project (201103013RC: RNA based gene testing using diagnostic minute samples for personalized therapy of lung cancer) will be used in the study.
* Patients have signed the informed consent (201103013RC) before 2019/01/31 and authorized the Institutional Review Board of Nation Taiwan University Hospital to review the new study for approving the usage of residual specimens.
* The residual samples from various sources, including surgical tissues, computed tomography (CT)-guided needle aspiration and/or biopsy, echo-guided needle aspiration and /or biopsy, bronchoscopic biopsy or brushing, bronchoalveolar lavage (BAL), endobronchial ultrasound guided needle aspiration, and lymph node aspiration, and pleural effusion specimens. The samples will be collected at the time of diagnostic procedure performed. All patients should sign an informed consent for purpose of using samples for molecular genetic testing.
* 600 residual specimens will be used for the study.

Exclusion Criteria:

* Patients didn't sign the informed consent (201103013RC).
* The residual specimens are not qualified.
* Patients didn't take epidermal growth factor receptor inhibitors.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: only citizens of Taiwan will be enrolled.
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Tumor size measurement for evaluating tumor progression | "up to 5 years," "from date of treatment (EGFR TKIs) until the date of first documented progression
  The change of tumor size is indicative of progression disease (PD) after EGFR TKI treatment.
  Tumor size is recorded using CT scan before the first day of of treatment and routine CT scan image is captured at each cycle of treatment to evaluate the growth of tumor.
  According to RECIST (The Response Evaluation Criteria in Solid Tumors), tumor progression will be assigned based on (1) a sum measurement of original target lesions that has increased more than 20%, (2) the reappearance of the original target lesions, (3) appearance of new lesions, and (4) a new lymph node metastatic lesion which is more than 10mm in diameter. Statistically, patients will be divided into two groups according to expression level of PTK7 mRNA, which is detected before the first dayof treatment. The clinicopathologic characteristics (sex, age, smoking history, EGFR mutation) will be enrolled in multivariate analysis.

SECONDARY OUTCOMES:
Lymph node lesion measurement for evaluating tumor metastasis | "up to 5 years," "from date of treatment (EGFR TKIs) until the date of first documented metastasis
  Lymph node metastatic lesion is recorded using CT scan before the first day of treatment and routine CT scan image is captured at each cycle of EGFR TKI treatment. A new lymph node metastatic lesion which is more than 10mm in diameter is considered as tumor metastasis.Statistically, patients will be divided into two groups according to expression level of PTK7 mRNA, which is detected before the first day of of treatment. The clinicopathologic characteristics (sex, age, smoking history, EGFR mutation) will be enrolled in multivariate analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Yuan Shih, Taipei, Taiwan